CLINICAL TRIAL: NCT07196501
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Maintenance of Effect of NBI-1065845 as an Adjunctive Treatment in Subjects With Major Depressive Disorder (MDD)
Brief Title: A Study to Evaluate the Maintenance Effect of NBI-1065845 as an Adjunctive Treatment in Participants With Major Depressive Disorder (MDD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1065845-MDD3027; 2025-520541-72-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; NBI-1065845
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study consists of a non-randomized open-label treatment period and a randomized double-blind maintenance period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open-label Treatment Period: NBI-1065845 (Experimental): Participants will be treated with NBI-1065845 during the open-label treatment period.
  Interventions: Drug: NBI-1065845
- Randomized Double-blind Maintenance Period: NBI-1065845 (Experimental): Participants will be randomized to receive NBI-1065845 during the randomized double-blind maintenance period.
  Interventions: Drug: NBI-1065845
- Randomized Double-blind Maintenance Period: Placebo (Experimental): Participants will be randomized to receive matching placebo during the randomized double-blind maintenance period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1065845 — Oral tablet
  Arms: Open-label Treatment Period: NBI-1065845; Randomized Double-blind Maintenance Period: NBI-1065845
Drug: Placebo — Oral tablet
  Arms: Randomized Double-blind Maintenance Period: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of NBI-1065845 compared with placebo as an adjunctive treatment in delaying relapse of depressive symptoms (maintenance of effect) in participants with MDD.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of recurrent MDD (moderate or severe) or persistent depressive disorder.
* Participant has had an inadequate response to oral antidepressant treatments in the current episode of depression.
* Participant must have been taking oral antidepressants for at least 8 weeks and is willing to continue the same oral antidepressants at the same dose and frequency of administration throughout participation in the study.
* Total Hamilton Depression Rating Scale-17 Item (HAM-D17) score ≥22 at screening and at study baseline (Day 1).
* Willing and able to comply with all study procedures and restrictions in the opinion of the investigator.

Key Exclusion Criteria:

* A current or prior psychiatric disorder diagnosis in the last 1 year that was the primary focus of treatment other than MDD.
* Are considered by the investigator to be at imminent risk of suicide or injury to self or others.
* Participants depressive symptoms have previously demonstrated nonresponse to electroconvulsive therapy (ECT) in the current major depressive episode.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Time from Randomization to Relapse | From randomization to the earliest of relapse or end-of study (up to approximately 32 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (28):
- United States (16):
  - Neurocrine Clinical Site, Oceanside, California
  - Neurocrine Clinical Site, New Haven, Connecticut
  - Neurocrine Clinical Site, Miami Gardens, Florida
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, Palm Bay, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, O'Fallon, Missouri
  - Neurocrine Clinical Site, Albuquerque, New Mexico
  - Neurocrine Clinical Site, Charlotte, North Carolina
  - Neurocrine Clinical Site, Edmond, Oklahoma
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Bellaire, Texas
  - Neurocrine Clinical Site, Friendswood, Texas
  - Neurocrine Clinical Site, Stafford, Texas
  - Neurocrine Clinical Site, Wichita Falls, Texas
  - Neurocrine Clinical Site, Draper, Utah
- Neurocrine Clinical Site, Sofia, Bulgaria
- Canada (3):
  - Neurocrine Clinical Site, North Vancouver, British Columbia
  - Neurocrine Clinical Site, Sherbrooke, Quebec
  - Neurocrine Clinical Site, Toronto
- Estonia (2):
  - Neurocrine Clinical Site, Tallinn
  - Neurocrine Clinical Site, Tartu
- Neurocrine Clinical Site, Rome, Italy
- Poland (3):
  - Neurocrine Clinical Site, Bialystok
  - Neurocrine Clinical Site, Bydgoszcz
  - Neurocrine Clinical Site, Gdansk
- Neurocrine Clinical Site, Barcelona, Spain
- Neurocrine Clinical Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No